CLINICAL TRIAL: NCT01281475
Title: A Phase 2 Randomized Placebo-Controlled Trial of Levodopa in Angelman Syndrome
Brief Title: A Trial of Levodopa in Angelman Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wen-Hann Tan (Other)
Collaborators: Rady Children's Hospital, San Diego (Other); University of California, San Francisco (Other); Baylor College of Medicine (Other); Vanderbilt University Medical Center (Other); Greenwood Genetic Center (Other); Children's Hospital Medical Center, Cincinnati (Other); Angelman Syndrome Foundation, Inc. (Other)
Responsible Party: Sponsor-Investigator, Wen-Hann Tan, Attending Physician in Genetics, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-12-0610; 3523 (Other Grant/Funding Number: OOPD)
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Angelman Syndrome
Keywords: Angelman syndrome; Levodopa; Carbidopa; L-dopa
MeSH Terms: conditions — Angelman Syndrome | interventions — Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levodopa (Experimental): Levodopa is prescribed as a combination of levodopa/carbidopa (4:1) to reduce the peripheral side effects. The dosage used was 15 mg/kg/day in 3 divided doses.
  Interventions: Drug: Levodopa
- Placebo (Placebo Comparator): The placebo contains excipients similar to those in the active drug, but it does not contain levodopa or carbidopa, so it is not expected to have any effect.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Levodopa — Levodopa/Carbidopa (4:1)
  Dosages are based on levodopa.
  Subjects randomized to the levodopa arm will receive a levodopa dose of 5 mg/kg/day in the first 2 weeks of the study, a levodopa dose of 10 mg/kg/day in the second 2 weeks of the study, and a levodopa dose of 15 mg/kg/day (up to a maximum of 800 mg per day) for the remaining duration of the study.
  Levodopa/Carbidopa is a combined formulation that will be dispensed as capsules. It should be taken 3 times a day.
  Other Names: Sinemet; L-dopa
  Arms: Levodopa
Drug: Placebo Oral Capsule — The placebo contains excipients similar to those in the active drug, but it does not contain levodopa or carbidopa.
  Arms: Placebo

SUMMARY:
This study is designed to determine whether levodopa will lead to an improvement in the development and tremor in children with Angelman syndrome (AS).

It has been suggested that levodopa, a medication that is usually used to treat Parkinson disease in adults, may help children with AS in their overall development and reduce the tremor that some of them have.

If levodopa is found to be beneficial for children with AS, this could lead to a new treatment for AS.

Funding Source - FDA-OOPD

DETAILED DESCRIPTION:
Levodopa is a prodrug that "delivers" dopamine to the brain. It is usually given with carbidopa, a peripheral decarboxylase inhibitor, to increase the bioavailability of levodopa. Animal studies have suggested that levodopa can reverse the excess phosphorylation of some enzymes involved in synaptic and neuronal function, including calcium/calmodulin-dependent kinase type 2 (CaMKII).

Recently, it was shown that excess phosphorylation of CaMKII may be responsible for some of the neurological deficits seen in Angelman syndrome. Therefore, it is hypothesized that levodopa may lead to an improvement in the neurodevelopment and abnormal movements (e.g. tremors) in children with Angelman syndrome.

Although many children have used levodopa for a variety of medical conditions over the last 30 years, it has not been approved by the Food and Drug Administration (FDA) for use in children, and it has not been formally studied in children with Angelman syndrome.

Therefore, the purpose of this study is to find out whether levodopa will lead to an improvement in the development and in the tremor in children with AS.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 4 years and 12 years (i.e., before the 13th birthday)
2. Molecular confirmation of the diagnosis of AS, which may include abnormal methylation studies or UBE3A mutation analyses - only subjects with a molecular diagnosis will be allowed to enroll
3. Not on LD, CD, or any dopamine agonists in the 2 weeks prior to participation

Exclusion Criteria:

1. Co-morbid disorders that may be associated with developmental or cognitive delays
2. Poorly controlled seizures - An average of more than 2 clinical seizures per month in the 12 months prior to enrollment.
3. Use of medications that may interact with LD/CD including atypical antipsychotics (aripiprazole, asenapine, iloperidone, olanzapine, paliperidone, risperidone, ziprasidone), monoamine oxidase inhibitors (isocarboxazid, phenelzine, selegiline, tranylcypromine), or phenytoin within the last 14 days, or other investigational interventions within the past 3 months
4. Presence of cardiovascular disease or instability, respiratory disease, liver disease, peptic ulcer disease, renal impairment, or hematological disorders
5. Pregnancy

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hann Tan, BMBS, Principal Investigator — Boston Children's Hospital; Lynne M. Bird, MD, Principal Investigator — Rady Children's Hospital, San Diego; Steven A. Skinner, MD, Principal Investigator — Greenwood Genetic Center; Carlos A. Bacino, MD, Principal Investigator — Baylor College of Medicine; Anne Slavotinek, MD, Principal Investigator — University of California, San Francisco; Cary Fu, MD, Principal Investigator — Vanderbilt University Medical Center; Logan Wink, M.D, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (7):
- United States (7):
  - Rady Children's Hospital, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Levodopa: Levodopa is a prodrug that "delivers" dopamine to the brain. It is usually given with carbidopa, a peripheral decarboxylase inhibitor, to increase the bioavailability of levodopa.
  Levodopa/carbidopa: Levodopa/Carbidopa (4:1)
  Dosages are based on levodopa.
  Subjects randomized to the levodopa arm will receive a levodopa dose of 5 mg/kg/day in the first 2 weeks of the study, a levodopa dose of 10 mg/kg/day in the second 2 weeks of the study, and a levodopa dose of 15 mg/kg/day (up to a maximum of 800 mg per day) for the remaining duration of the study.
  Levodopa/Carbidopa is a combined formulation that will be dispensed as capsules. It should be taken 3 times a day.
- Placebo: The placebo (in this study, microcellulose) is not expected to have any effect.
Period: Overall Study
Arm/Group | Levodopa | Placebo
Started | 33 | 34
Completed | 29 | 26
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study were analyzed. Therefore all numbers in the Results section refer to the participants who completed the study.
Groups:
- Placebo: The placebo (in this study, microcellulose) is not expected to have any effect.
  It is also taken 3 times a day, just like Levodopa.
- Total: Total of all reporting groups
Arm/Group | Levodopa | Placebo | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Categorical [Count of Participants; unit: Participants] — In the Levodopa group, 4 participants failed to complete the study; in the Placebo group, 8 participants failed to complete the study. None of these 12 participants could be analyzed further, so we do not have the breakdown of their gender and other measures.
  Participants
    <=18 years | 29 | 26 | 55
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 13 | 12 | 25
  Male | 16 | 14 | 30
Developmental age - Bayley Cognitive [Mean (Standard Deviation); unit: months] | 19 (8) | 18 (6) | 19 (7)
Tremors [Count of Participants; unit: Participants] — Presence of tremors at baseline
  Participants | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Bayley Cognitive Age Equivalent at 1 Year
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: months
Groups:
- Placebo: The placebo (in this study, microcellulose) is not expected to have any effect.
  The placebo capsules are taken 3 times a day, just like the levodopa / carbidopa capsules
Arm/Group | Levodopa | Placebo
Number analyzed (Participants) | 29 | 26
months | 19 (7) | 19 (8)
Statistical Analysis 1: Comparison: Levodopa vs Placebo; We performed generalized estimating equations with an unstructured covariance matrix to account for inter-correlations within measurements on the same participant over time; Test type: Superiority — We modeled each outcome variable as a function of treatment (ie, levodopa versus placebo), visit (ie, baseline vs. 12-month follow-up) and the treatment-by-visit interaction; the interaction term tests whether the effect of levodopa treatment over time is significantly greater than that of the placebo group; p = 0.75, Generalized estimating equations — This was the calculated p value without correction for multiple comparisons

2. Secondary Outcome: Presence of Tremors
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Levodopa: Levodopa is prescribed as a combination of levodopa/carbidopa (4:1) to reduce the peripheral side effects. The dosage used was 15 mg/kg/day in 3 divided doses.
  Levodopa: Levodopa/Carbidopa (4:1)
  Dosages are based on levodopa.
  Subjects randomized to the levodopa arm will receive a levodopa dose of 5 mg/kg/day in the first 2 weeks of the study, a levodopa dose of 10 mg/kg/day in the second 2 weeks of the study, and a levodopa dose of 15 mg/kg/day (up to a maximum of 800 mg per day) for the remaining duration of the study.
  Levodopa/Carbidopa is a combined formulation that will be dispensed as capsules. It should be taken 3 times a day.
Arm/Group | Levodopa | Placebo
Number analyzed (Participants) | 29 | 26
Participants | 14 | 12

ADVERSE EVENTS:
Arm/Group | Levodopa | Placebo
Serious Adverse Events (participants affected / at risk) | 3/33 | 1/34
Other Adverse Events (participants affected / at risk) | 11/33 | 9/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa (N=33) | Placebo (N=34)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa (N=33) | Placebo (N=34)
Seizures (Nervous system disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No